CLINICAL TRIAL: NCT05030974
Title: Optimal Repeated Dose Strategy for SARS-CoV-2 Vaccination in Kidney Transplant Patients A Prospective, Randomized Multicenter Study by the REnal Patients COVID-19 VACcination (RECOVAC) Consortium
Brief Title: RECOVAC Repeated Vaccination Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other); Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL78963.042.21
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Kidney Diseases; Vaccine Response Impaired; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19; Kidney Diseases | interventions — 2019-nCoV Vaccine mRNA-1273; Ad26COVS1

STUDY DESIGN:
Intervention Model Description: Based on their immunosuppressive treatment, patients will participate in one of the following strata:
  * stratum A: patients treated with triple immunosuppressive therapy consisting of a calcineurin inhibitor, MMF/MPA, and steroids,
  * stratum B: patients treated with any combination of immunosuppressive drugs.
  In stratum A, patients will be randomized to one of two third or fourth vaccination strategies:
  * A1: one extra dose of mRNA-1273 (100 μg, i.m)
  * A2: one extra dose of mRNA-1273 (100 μg, i.m), with temporary discontinuation of MMF/MPA during one week before and one week after the 3rd dose
  In stratum B, patients will be randomized to one of three third vaccination strategies:
  * B1: 3rd dose of mRNA-1273 (100 μg, i.m)
  * B2: 3rd dose of mRNA-1273 (100 μg, i.m) in both upper arms
  * B3: Ad26.COV2.S vaccine (Janssen, 5x1010 viral particles i.m.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- stratum A1 - one extra dose of mRNA-1273 (Active Comparator): Patients treated with triple immunosuppressive therapy consisting of a calcineurin inhibitor, MMF/MPA, and steroids, receiving a 3rd or 4th dose of mRNA-1273 (100 μg, i.m)
  Interventions: Biological: mRNA-1273
- stratum A2 - one extra dose of mRNA-1273 with discontinuation of MMF/MPA (Active Comparator): patients treated with triple immunosuppressive therapy consisting of a calcineurin inhibitor, MMF/MPA, and steroids, receiving a 3rd or 4th dose of mRNA-1273 (100 μg, i.m), with temporary discontinuation of MMF/MPA during one week before and one week after the extra dose
  Interventions: Biological: mRNA-1273
- stratum B1 - 3rd dose of mRNA-1273 (Active Comparator): patients treated with any combination of immunosuppressive drugs, receiving a 3rd dose of mRNA-1273 (100 μg, i.m)
  Interventions: Biological: mRNA-1273
- statum B2 - 3rd double dose of mRNA-1273 (Active Comparator): patients treated with any combination of immunosuppressive drugs, receiving a 3rd dose of mRNA-1273 (100 μg, i.m) in both upper arms
  Interventions: Biological: mRNA-1273
- stratum B3 - Ad26.COV2.S vaccine (Active Comparator): patients treated with any combination of immunosuppressive drugs, receiving a 3rd COVID vaccination with Ad26.COV2.S vaccine (Janssen, 5x1010 viral particles i.m.)
  Interventions: Biological: Ad26.COV2.S vaccine

INTERVENTIONS:
Biological: mRNA-1273 — SARS-CoV-2 vaccination
  Arms: statum B2 - 3rd double dose of mRNA-1273; stratum A1 - one extra dose of mRNA-1273; stratum A2 - one extra dose of mRNA-1273 with discontinuation of MMF/MPA; stratum B1 - 3rd dose of mRNA-1273
Biological: Ad26.COV2.S vaccine — SARS-CoV-2 vaccination
  Arms: stratum B3 - Ad26.COV2.S vaccine

SUMMARY:
Rationale: The humoral and cellular immune response after two mRNA vaccinations is severely attenuated in kidney transplant patients compared to controls, especially when their immunosuppressive regimen contains mycophenolate mofetil (MMF) / mycophenolic acid (MPA). A repeated dose strategy is therefore required to improve the efficacy of vaccination.

Objective: To investigate the immunogenicity of third or fourth dose SARS-CoV-2 vaccination strategies in kidney transplant patients.

Study design: Prospective, multicentre, open-label randomized clinical trial

Study population: Patients with a functioning kidney transplant who did not seroconvert after two or three doses of a mRNA vaccine (either mRNA-1273 (Moderna) or BNT162b2 (Pfizer) or any combination of both)

Procedures:

Based on their immunosuppressive treatment, patients can participate in one of the following strata:

* stratum A: patients receiving triple immunosuppressive therapy, consisting of a calcineurin inhibitor, MMF/MPA, and steroids In stratum A, patients will be randomized to one of two equally sized groups. Patients will receive a third or fourth vaccination of the mRNA-1273 vaccine (100 μg, i.m), with either continuation of MMF/MPA (A1) or discontinuation of MMF/MPA during one week before and one week after the third or fourth dose, respectively (A2).
* stratum B: patients receiving any combination of immunosuppressive drugs. In stratum B, patients will be randomized to one of three equally sized groups. Patients will receive another dose (100 μg, i.m) of the mRNA-1273 vaccine (B1), or two single doses of mRNA-1273 into the left and the right upper arm (2 x 100 μg, i.m; B2), or the Ad26.COV2.S vaccine (Janssen, 5x1010 viral particles, i.m; B3).

Main study parameters/endpoints:

The primary endpoint is the proportion of patients with an anti-S1 antibody concentration higher than 10 BAU/mL established at 28 days after the third or fourth vaccine administration. Within each stratum different vaccination strategies will be compared.

Secondary endpoints include:

* concentration of anti-S1 antibodies in serum at 28 days after the 3rd or 4th vaccine administration
* concentration of virus-neutralizing antibodies in serum
* SARS-CoV-2 specific T cell responses
* safety in terms of incidence of acute rejection and solicited local and systemic adverse events (AEs) after vaccination.
* antibody (IgG and IgA) responses in nasal mucosal fluid

DETAILED DESCRIPTION:
2. OBJECTIVES

Primary objective:

To assess the immunogenicity (expressed as percentage of responders) of various COVID-19 third or fourth vaccination strategies in kidney transplant patients that failed to mount a sufficient antibody response after two or three primary doses of a mRNA vaccine (either mRNA-1273 (Moderna) or BNT162b2 (Pfizer) or any combination of both).

Secondary Objectives:

* To measure the concentration of SARS-CoV-2 spike S1-specific IgG antibodies in serum at 28 days after the 3rd or 4th vaccine administration
* To measure the presence and titer of neutralizing anti-SARS-CoV-2 antibodies after third or fourth vaccination
* To evaluate SARS-CoV-2 specific T cell responses
* To measure anti-S1 antibody (IgG and IgA) responses and neutralizing capacity of these antibodies in nasal mucosal fluid
* To evaluate vaccine safety in terms of incidence of solicited local and systemic adverse events (AEs) graded according to severity.

Exploratory Objectives:

* To assess the association between baseline clinical and immunological parameters and the immune response to third or fourth vaccinations
* To correlate RNA-seq data at one week after vaccination to the subsequent antibody and T cell response

  3. STUDY DESIGN

This is a prospective, multicentre, open-label, randomized study to evaluate the immunogenicity and safety of various third or fourth vaccination strategies in kidney transplant patients without a sufficient antibody response after two or three primary doses of a mRNA vaccine (either mRNA-1273 (Moderna) or BNT162b2 (Pfizer) or any combination of both).

The four participating study sites are: Amsterdam UMC, ErasmusMC, Radboudumc and UMCG.

Based on their immunosuppressive treatment, patients will participate in one of the following strata:

* stratum A: patients treated with triple immunosuppressive therapy consisting of a calcineurin inhibitor, MMF/MPA, and steroids,
* stratum B: patients treated with any combination of immunosuppressive drugs.

In stratum A, patients will be randomized to one of two third or fourth vaccination strategies:

* A1: one extra dose of mRNA-1273 (100 μg, i.m)
* A2: one extra dose of mRNA-1273 (100 μg, i.m), with temporary discontinuation of MMF/MPA during one week before and one week after the 3rd dose

In stratum B, patients will be randomized to one of three third vaccination strategies:

* B1: 3rd dose of mRNA-1273 (100 μg, i.m)
* B2: 3rd dose of mRNA-1273 (100 μg, i.m) in both upper arms
* B3: Ad26.COV2.S vaccine (Janssen, 5x1010 viral particles i.m.)

To assess the immune response after vaccination, blood samples will be collected at baseline (i.e. prior to third dose administration) and at 28 days after the third or fourth dose administration. A complete blood count, kidney function, and liver enzymes will be determined at the same time points.

In a subset of patients we will collect a blood sample at 1 week after the third vaccin administration for specific immunological assays.

For safety reasons, a blood sample will be collected in stratum A at one and two weeks after discontinuing MMF/MPA.

The maximum volume of blood collected for this study is 66 mL per timepoint, and no more than 200 mL for the one year study period, which is well within the safe limits of blood collection for clinical studies.

Nasal mucosal lining fluid (MLF) will be collected for assessment of secreted mucosal antibodies at the same time points used to collect blood. MLF will be collected by use of soft synthetic absorptive matrix (SAM) strips, which are gently inserted into one nostril of the participant and placed along the surface of the inferior turbinate. The index finger is then lightly pressed against the side of the nostril to keep the SAM strip in place and to allow MLF absorption for 60 seconds, after which the SAM strip is placed back in the protective plastic tube. The procedure may tickle slightly but is completely painless.

To evaluate vaccination related AEs, patients will be asked to collect solicited local and systemic AEs for 7 days after each vaccination using a questionnaire, as vaccination related AEs are mainly expected in the first week after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Received 2 doses of mRNA-1273 (stratum B) according to the recommended vaccination schedule, with the last administration within the last nine months. For stratum A, also patients who received 2 doses of BNT162b2 and/or a third dose with a mRNA vaccine (mRNA-1273 or BNT162b2) within the last three months are eligible.
3. At least 6 months after kidney transplantation
4. Negative seroresponse 14 to 56 days after vaccination, measured by a validated anti-spike IgG assay of which the definition is dependent on the assay that is used.
5. Eligible for COVID-19 vaccination as described by the instructions of the manufacturers of the vaccine (Moderna and Janssen)
6. Capable of understanding the purpose and risks of the study, fully informed and given written informed consent (signed informed consent form has been obtained)
7. Willing to adhere to the protocol and be available during the study period

   Additional inclusion criteria to be eligible for stratum A:
8. Maintenance immunosuppressive therapy consisting of a calcineurin inhibitor (tacrolimus or cyclosporine), MMF/MPA, and prednisone
9. In case of tacrolimus treatment: last tacrolimus pre-dose level while on current dosage above 4 μg/l
10. In case of cyclosporine treatment: last cyclosporine pre-dose level while on current dosage above 75 μg/l
11. Prednisone dose at least 5 mg/day
12. First or second transplantation
13. Calculated level of panel reactive antibodies prior to last transplantation below 85%
14. No signs of acute rejection during the preceding year

Exclusion Criteria:

1. Multi-organ transplant recipient
2. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s).
3. Previous or active COVID-19 disease
4. Active malignancy, except non-melanoma skin cancer
5. Inherited immune deficiency
6. Infection with Human Immunodeficiency Virus (HIV)
7. Administration of T cell, B cell, or plasma cell depleting antibodies during the last 6 months
8. Any vaccination within a week before enrolment
9. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.

   Additional exclusion criteria for stratum B:
10. History of recurrent venous thrombosis or venous thrombosis <2 years before baseline
11. Immune-mediated diseases associated with thrombocytopenia such as ITP and aHUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Positive SARS-CoV-2 seroresponse | 28 days after third vaccination
  The percentage of subjects with a serum anti-S1 IgG concentration ≥10 BAU/mL after the third or fourth vaccine administration

SECONDARY OUTCOMES:
SARS-CoV-2 antibody concentration | 28 days after vaccination
  SARS-CoV-2 anti-S1 IgG concentration in serum after third or fourth vaccine administration
Virus-neutralizing capacity of SARS-CoV-2 antibodies | 28 days after vaccination
  The titer of neutralizing anti-SARS-CoV-2 antibodies after third or fourth vaccine administration
Mucosal SARS-CoV-2 antibodies | 28 days after vaccination
  Concentrations of SARS-CoV-2 specific antibodies (IgG and IgA) in nasal fluid after third or fourth vaccine administration
SARS-CoV-2 specific T cell response | 28 days after vaccination
  1. Interferon-gamma concentration in whole blood after ex vivo stimulation with SARS-CoV-2 specific peptides
  2. Ex vivo production of T cell related cytokines by peripheral blood mononuclear cells (PBMC) in ELISpot assays after third vaccine administration
Solicited local and systemic adverse events | within 7 days after vaccination
  Percentage of participants reporting local reactions (pain at the injection site, redness and swelling) and systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new of worsened muscle pain, and new or worsened joint pain) after third or fourth vaccine administration
Serious adverse events | within 28 days after vaccination
  Percentage of participants with serious adverse events after third or fourth vaccine administration

OTHER OUTCOMES:
Relation between age and immune response | 28 days after vaccination
  The association between age and development of an antibody and/or T cell response after third or fourth vaccine administration
Relationship between time after transplant and immune response | 28 days after vaccination
  The association between time after transplantation and development of an antibody and/or T cell response after third or fourth vaccine administration
Relationship between immunosuppressive medication and immune response | 28 days after vaccination
  The association between baseline immunosuppressive medication and development of an antibody and/or T cell response after third or fourth vaccine administration
Relationship between lymphocytes and immune response | 28 days after vaccination
  The association between baseline lymphocytes and development of an antibody and/or T cell response after third or fourth vaccine administration
Relationship between eGFR and immune response | 28 days after vaccination
  The association between baseline eGFR and development of an antibody and/or T cell response after third or fourth vaccine administration
SARS-CoV-2 reactive CD4+ and CD8+ cells | 28 days after vaccination
  Flow cytometry of PBMC for measuring SARS-CoV-2 reactive CD4+ and CD8+ cells after third or fourth vaccine administration
Early gene expression for SARS-CoV-2 immune response | 28 days after vaccination
  RNA-seq analysis to detect early gene expression that are associated with the development of an antibody and/or T cell response after third or fourth vaccine administration
Incidence of COVID-19 breakthrough infection | 28 days after vaccination
  Measured by questionnaires and SARS-CoV-2 nucleocapsid specific antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan F Sanders, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (4):
  - Radboud umc, Nijmegen, Gelderland
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus mc, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: No
The data of this study will be available from the principal investigator, upon reasonable request.

REFERENCES:
- [Derived] Vervoort JPM, Konijn WS, Jansen DEMC, Boersma C, de Zeeuw J, Ho-Dac-Pannekeet MM, Gansevoort RT, Messchendorp AL, Sanders JSF, de Wildt-Liesveld R. Patient engagement as a collaborative process in a large Dutch COVID-19 vaccination study (RECOVAC) - insight into the contribution of patient engagement and learnings for the future. Res Involv Engagem. 2024 Sep 13;10(1):96. doi: 10.1186/s40900-024-00622-x. PMID 39272117
- [Derived] Malahe SRK, den Hartog Y, Rietdijk WJR, van Baarle D, de Kuiper R, Reijerkerk D, Ras AM, Geers D, Diavatopoulos DA, Messchendorp AL, van der Molen RG, Imhof C, Frolke SC, Bemelman FJ, Gansevoort RT, Hilbrands LB, Sanders JF, GeurtsvanKessel CH, Kho MML, de Vries RD, Reinders MEJ, Baan CC; On behalf of RECOVAC Consortium. Repeated COVID-19 Vaccination Drives Memory T- and B-cell Responses in Kidney Transplant Recipients: Results From a Multicenter Randomized Controlled Trial. Transplantation. 2024 Dec 1;108(12):2420-2433. doi: 10.1097/TP.0000000000005119. Epub 2024 Nov 21. PMID 38902860
- [Derived] Kho MML, Messchendorp AL, Frolke SC, Imhof C, Koomen VJ, Malahe SRK, Vart P, Geers D, de Vries RD, GeurtsvanKessel CH, Baan CC, van der Molen RG, Diavatopoulos DA, Remmerswaal EBM, van Baarle D, van Binnendijk R, den Hartog G, de Vries APJ, Gansevoort RT, Bemelman FJ, Reinders MEJ, Sanders JF, Hilbrands LB; RECOVAC collaborators. Alternative strategies to increase the immunogenicity of COVID-19 vaccines in kidney transplant recipients not responding to two or three doses of an mRNA vaccine (RECOVAC): a randomised clinical trial. Lancet Infect Dis. 2023 Mar;23(3):307-319. doi: 10.1016/S1473-3099(22)00650-8. Epub 2022 Oct 27. PMID 36354032